CLINICAL TRIAL: NCT00927797
Title: Phase II Study to Evaluate the Safety and Efficacy of the Treatment With Pentostatin, Cyclophosphamide and Rituximab Followed by Rituximab Maintenance in Previously Untreated and Relapsed Patients With Immunocytoma/Morbus Waldenström, B-CLL and Other Indolent B-Cell Lymphomas
Brief Title: Interventional Study on Pentostatin, Cyclophosphamide and Rituximab in Indolent B-Cell Non-Hodgkin-Lymphoma (B-NHL)
Acronym: PERLL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Diakonie Krankenhaus Schwäbisch Hall, Germany (Unknown); Ludwig-Maximilians - University of Munich (Other); Klinikum am Plattenwald, Bad Friedrichshall, Germany (Unknown); Diakonie-Klinikum Stuttgart (Other); Gemeinschaftspraxis Porowski & Koniczek, Heilbronn, Germany (Unknown); Universitätsmedizin Mannheim (Other)
Responsible Party: Prof. Dr. med. A. D. Ho, University of Heidelberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-278/2004; BfArM 4022892
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Immunocytoma/Morbus Waldenström; B-Cell Non-Hodgkin's Lymphoma; B-Cell Chronic Lymphocytic Leukemia
Keywords: immunochemotherapy; Pentostatin; Cyclophosphamide; Rituximab; Maintenance; indolent B-NHL; B-CLL; B-NHL
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; Pentostatin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunochemotherapy, Maintencance (Experimental)
  Interventions: Drug: Cyclophosphamide, Pentostatin, Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide, Pentostatin, Rituximab

SUMMARY:
The combination of Fludarabine and Cyclophosphamide have yielded overall response rates of over 80% in previously untreated patients with indolent Non-Hodgkin-Lymphoma. However, hematotoxicity rates were high with Grade 3 and 4 toxicities of over 50%. Several studies have indicated that the treatment with Pentostatin and Cyclophosphamide causes lower hematotoxicity rates than the combination of Fludarabine and Cyclophosphamide. To evaluate the efficacy and safety of treatment with Pentostatin/Cyclophosphamide immuno-chemotherapy for patients with newly diagnosed or relapsed Immunocytoma/Morbus Waldenström, B-cell chronic lymphocytic leukemia (B-CLL) and other indolent CD20-positive B-NHL, an open, non-randomized, multi-center prospective phase II-study to evaluate the efficacy and safety of treatment with immuno-chemotherapy is conducted. Treatment consists of 6 courses of Pentostatin (4mg/m² on day 1), Cyclophosphamide (600mg/m² on day 1) and Rituximab (375mg/m² on day 0) administered every three weeks. Patients achieving complete or partial remission undergo maintenance therapy consisting of 8 courses of Rituximab (375mg/m²) administered every three months over a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* confirmed first diagnosis of or relapsed CD20-positive Immunocytoma, B-CLL or other indolent B-NHL
* therapy-requiring CLL defined as: Binet stage C or Binet B combined with occurence of B-symptoms, rapidly progressing disease, risk of organ compression by lymphoma mass
* therapy-requiring Immunocytoma as defined by the Consensus Panel Recommendations from the Second International Workshop on Waldenström´s Macroglobulinemia, 2003)
* age > 18 years
* anticipated life expectancy > 6 months
* ECOG 0-3
* no significant comorbidities
* signed informed consent
* efficient method of contraception during time of therapy (men and women)

Exclusion Criteria:

* age < 18 years
* CD20 negativity
* significant comorbidities interfering with therapy as required by the protocol
* history of HIV infection or active hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2005-02; Primary Completion 2009-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: overall response rate | after 6 months and after 36 months

SECONDARY OUTCOMES:
Toxicity according to WHO-Grading | throughout the treatment and until 36 months after
Efficacy: complete remission rate | after 6 months and 36 months
Efficacy: partial remission rate | after 6 months and 36 months
Efficacy: progression-free survival | after 6 months and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Ho, Ph.D., Prof., Principal Investigator — Director of Department

REFERENCES:
- See also: Homepage of the Department — http://www.klinikum.uni-heidelberg.de